CLINICAL TRIAL: NCT06559462
Title: Optimizing Nudge Strategies to Increase the Adoption of DPYD Testing in Patients With Gastrointestinal (GI) Malignancies Treated With Fluoropyrimidines.
Brief Title: Nudge Strategies for DPYD Testing in Patients With Gastrointestinal Cancers Treated With Fluoropyrimidines
Acronym: DPYD Nudges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UPCC 05224
Record Dates: First submitted 2024-07-25; First posted 2024-08-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: DPYD Gene Mutation; Gastrointestinal Cancer; Health Care Seeking Behavior
Keywords: Pharmacogenomic Testing; Pharmacogenetic Testing; Nudges; Implementation
MeSH Terms: conditions — Gastrointestinal Neoplasms; Patient Acceptance of Health Care | interventions — Focus Groups

STUDY DESIGN:
Intervention Model Description: Patients and providers will either participate in focus groups or complete a survey to provide feedback on developing nudges
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Physician Focus Group (Other): To develop patient- and clinician-directed nudges that will address biases to DPYD testing. Clinicians will be engaged to provide input on developing the content and design of the nudges that address biases that impact the decision to order DPYD testing. Feedback will be elicited for nudges based on relevancy, nudge timing, and appropriateness. We will also develop/refine patient- and clinician-focused educational materials and test results based on input from our focus groups.
  Interventions: Other: Focus Group
- Patient Focus Group (Other): To develop patient-directed nudges that will address biases to DPYD testing. Patients will be engaged to provide input on developing the content and design of the nudges that address biases that impact the decision to order DPYD testing. Feedback will be elicited for nudge content, clarity, and perceived urgency. We will also develop/refine patient-focused educational materials and test results based on input from our focus groups.
  Interventions: Other: Focus Group
- Physician Discrete Choice (Experimental): To pilot test clinician-nudges using discrete choice experiments, we will test the degree each nudge is associated with the perceived intention to order testing (clinician). Clinicians will be shown a series of nudges, and asked to choose which of each pair is the better nudge. The location/timing of the nudge in their workflow will be presented as part of the discrete choice.
  Interventions: Other: Discrete Choice
- Patient Discrete Choice (Experimental): To pilot test patient-nudges using discrete choice experiments, we will test the degree each nudge is associated with perceived likelihood to prompt discussion regarding testing. Patients will be shown a series of nudges, and asked to choose which of each pair is the better nudge.
  Interventions: Other: Discrete Choice

INTERVENTIONS:
Other: Focus Group — Open-ended group discussion of potential nudges to elicit constructive feedback on nudge development.
  Arms: Patient Focus Group; Physician Focus Group
Other: Discrete Choice — Survey involving choice between two potential nudges to elicit feedback on which nudge version is considered superior.
  Arms: Patient Discrete Choice; Physician Discrete Choice

SUMMARY:
5-fluorouracil and capecitabine, sometimes called 5-FU, fluoropyrimidines, or Xeloda are a type of chemotherapy. Many people have side effects from these drugs like nausea, diarrhea, or blood problems. This research study is being conducted to learn how to help increase the number of patients offered DPYD testing before taking this type of chemotherapy drugs. DPYD testing can help predict risk of side effects.

Different people's bodies break down and use drugs faster or slower. Genes are the instructions that tell our bodies how to do this. The DPYD gene is one of the genes that tell your body how to use chemotherapy drugs. Some people have changes in their DPYD gene that can make their side effects from chemotherapy worse, sometimes so bad that they die. DPYD testing can tell doctors which people have these gene changes and need extra monitoring during chemotherapy.

Some of the people in this study will join a focus group and read sample messages for future patients. They will discuss with the other participants how well the message does its job and anything that might make the message better. When there are no more messages, the host may ask about other information for future patients like a website or brochure.

Other people in the study will read sample messages that may be sent to future patients about DPYD testing. They will select the message that they like the best and might make them ask their oncologist about testing options.

DETAILED DESCRIPTION:
INTRODUCTION AND PURPOSE:

Fluoropyrimidines (FPs) are the cornerstone of treatment for several gastrointestinal (GI) malignancies. Approximately 5-7% of patients carry reduced function variants in DPYD, resulting in the inability to metabolize FPs, predisposing them to severe, life-threatening toxicities. These patients can be identified through DPYD pharmacogenetic (PGx) testing. However, DPYD testing has not been widely adopted in clinical care due to implementation barriers at the system- (e.g., access to testing, integration into clinical workflows), clinician- (e.g., interpretation of results, remembering to order test) and patient- (e.g., knowledge about testing, worry about adverse effects of testing) levels. This results in substantial uncertainty and a tendency to rely on several biases [e.g., status quo (not to test), loss aversion (perception of loss greater than gain), omission (focusing on harm of action more than of non-action), or confirmation (validating prior beliefs)] that can influence health decisions. Behavioral economics offers a roadmap for mitigating clinician biases using choice architecture and message framing, which involves changing the EHR environment to facilitate the desired (evidence-based) choice, and patient biases using priming, which uses direct communication strategies to address potential biases prior to clinical encounters. In Aim 1, we will develop patient- and clinician-directed nudges with input from key stakeholders. Feedback will also be used to develop and refine educational materials to support clinical testing. In Aim 2, we will pilot test the nudges using discrete choice experiments (DCE) to identify the optimal framing that best mitigate cognitive biases. Results of the pilot will be utilized to design a randomized clinical trial testing the nudge strategies.

OBJECTIVES:

To obtain input from clinician and patient stakeholders to design EHR based nudges that are acceptable and will increase the likelihood of ordering DPYD testing prior to prescribing a FP for GI cancer.

Aim 1: Develop and refine patient- and clinician- directed nudges that will address biases to DPYD testing. Hypothesis: Stakeholder feedback will result in acceptable and appropriate nudges.

Aim 1a. We will conduct focus groups with stakeholders and clinicians to refine the framing and content of EHR nudges that will best mitigate biases to ordering DPYD testing.

Aim 1b. We will conduct focus groups with patients to refine the framing of patient directed nudges that would prompt them to initiate discussion about DPYD testing with clinicians.

Aim 1c. Feedback from stakeholders will also be used to develop/refine clinician and patient educational websites.

Aim 2: Pilot test patient- and clinician- nudges using discrete choice experiments.

We will test the degree to each message is associated with the greatest intention to order testing (clinician), or prompt discussion regarding testing (patient) with in a sample of 35 clinicians and 75 patients.

The results of this pilot will be used as preliminary data for a NIH grant to conduct a prospective randomized, implementation trial to evaluate the effectiveness of the optimized nudges to enhance the adoption of DPYD testing as an evidence-based way to reduce TRAEs and improve the quality of care for cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Currently involved in the practice or policy of GI oncology/DPYD testing/FP use/Healthcare Development OR
* Prescribed a FP for GI cancer diagnosis in the past six months AND Currently licensed to provide health care in Pennsylvania or New Jersey OR
* Previous diagnosis of GI malignancy or family member who had GI malignancy

Exclusion Criteria:

* Less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Developmental Nudge Feedback | 90 minutes
  Verbal data collected and coded
Discrete Nudge Feedback | 45 minutes
  Binary choices

CONTACTS AND LOCATIONS:
Overall Officials: Sony Tuteja, PharmD, MS, Principal Investigator — Abramson Cancer Center
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lau-Min KS, Varughese LA, Nelson MN, Cambareri C, Reddy NJ, Oyer RA, Teitelbaum UR, Tuteja S. Preemptive pharmacogenetic testing to guide chemotherapy dosing in patients with gastrointestinal malignancies: a qualitative study of barriers to implementation. BMC Cancer. 2022 Jan 8;22(1):47. doi: 10.1186/s12885-022-09171-6. PMID 34996412
- [Background] Varughese LA, Bhupathiraju M, Hoffecker G, Terek S, Harr M, Hakonarson H, Cambareri C, Marini J, Landgraf J, Chen J, Kanter G, Lau-Min KS, Massa RC, Damjanov N, Reddy NJ, Oyer RA, Teitelbaum UR, Tuteja S. Implementing Pharmacogenetic Testing in Gastrointestinal Cancers (IMPACT-GI): Study Protocol for a Pragmatic Implementation Trial for Establishing DPYD and UGT1A1 Screening to Guide Chemotherapy Dosing. Front Oncol. 2022 Jul 5;12:859846. doi: 10.3389/fonc.2022.859846. eCollection 2022. PMID 35865463
- [Background] Hoffecker G, Varughese LA, Bleznuck J, Landgraf J, Wollack C, Chen J, Ritchie MD, Nathanson KL, Tuteja S. Customizing the electronic health record for delivery of pharmacogenetics. Genet Med Open. 2023 Mar 8;1(1):100779. doi: 10.1016/j.gimo.2023.100779. eCollection 2023. No abstract available. PMID 39669236